CLINICAL TRIAL: NCT00399477
Title: Open-label, Multicenter, Effectiveness and Safety Study of Once Daily AZILECT® as Mono- or Adjunct Therapy in Patients With Idiopathic Parkinson's Disease (PD)
Brief Title: A Non-Blinded Study Demonstrating the Effectiveness and Safety of Azilect Alone or in Combination Therapy in Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Neuroscience, Inc. (Industry)
Responsible Party: Thomas Smith, MD, Teva Neuroscience
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TVP-1012/PM101
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline; Pramipexole; Levodopa; ropinirole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rasagiline mesylate (Active Comparator)
  Interventions: Drug: rasagiline mesylate
- Rasagiline mesylate plus adjunct therapy (Experimental): Rasagiline mesylate with one of three adjunct therapies
  Interventions: Drug: Rasagiline mesylate plus Mirapex; Drug: Rasagiline mesylate with Levodopa; Drug: Rasagiline mesylate with Requip

INTERVENTIONS:
Drug: rasagiline mesylate — Azilect®
  Arms: Rasagiline mesylate
Drug: Rasagiline mesylate plus Mirapex — Mirapex, Azilect®
  Arms: Rasagiline mesylate plus adjunct therapy
Drug: Rasagiline mesylate with Levodopa — Azilect®, Levodopa
  Arms: Rasagiline mesylate plus adjunct therapy
Drug: Rasagiline mesylate with Requip — Azilect®, Requip
  Arms: Rasagiline mesylate plus adjunct therapy

SUMMARY:
Patients with Parkinson's Disease (PD) will be divided into 2 groups at each study center at their first visit based on the drugs they are taking for their PD:

* Group 1 Patients using Azilect and no other therapy.
* Group 2 Azilect in combination with other medications like Levodopa, Mirapex, or Requip.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic Parkinson's disease. Diagnosis previously confirmed by the presence of bradykinesia and by at least one additional cardinal sign (i.e., resting tremor, rigidity), without other known or suspected cause of parkinsonism.
2. Requiring therapy for PD symptom control

   * Azilect monotherapy.
   * Azilect as adjunct therapy..

Exclusion Criteria:

1. Patients previously exposed to Azilect
2. Patients with pheochromocytoma
3. Concomitant MAO inhibitors or medications contraindicated for use with MAO inhibitors are not allowed.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To identify the earliest scheduled visit of symptomatic effect | 8 months

SECONDARY OUTCOMES:
To characterize the effectiveness of Azilect in a usual community neurological | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: MerriKay Oleen-Burkey, PhD, Study Director — Teva Neuroscience, Inc.